CLINICAL TRIAL: NCT04787770
Title: The Role of HSP90 in Peripheral Vascular Lesions of Diabetic Atherosclerosis
Acronym: rhsppvlda
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-268
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease
Keywords: diabetic disease; peripheral arterial disease; Extracellular heat shock protein 90
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diabetes without complications: diabetes without complications
  Interventions: Other: non-intervention
- diabetes with Peripheral Arterial Disease: diabetes with Peripheral Arterial Disease
  Interventions: Other: non-intervention
- diabetic foot group: diabetic foot group
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
Diabetic foot disease with a global incidence of about 6% is one of the most serious complications of diabetes, which brings great pain and economic burden to patients.In China, the incidence rate is 8.1%, and the amputation rate is 7.3%. Every year, more than 1 million diabetic patients have amputations, ranking first among non-traumatic amputations.According to the American Diabetes Association (ADA), the incidence of Peripheral Arterial Disease (PAD) in diabetic patients is twice that of non-diabetic patients, and the resulting lower limb ischemia is the main cause of the high mortality and disability rate of diabetic foot.According to the International Working Group on Diabetic Foot (IWGDF), about 50% patients with diabetic foot disease are complicated with PAD, and the degree of vascular stenosis is closely related to the prognosis.Severe limb ischemia is a higher cause of diabetic foot ulcer in China than in western countries.Atherosclerosis is the main pathological change of diabetic peripheral artery disease, and endothelial injury is the initial link of atherosclerosis.Heat shock protein 90 (HSP90) is a kind of important heat stress protein, which accounts for about 2-3% of the total protein in cells.It is involved in the correct folding and activation of intracellular proteins.Although Hsp90 is primarily involved in intracellular protective mechanisms, they can also be exposed to the plasma membrane and released in the extracellular space, resulting in detectable levels of Hsp90 in the blood.Extracellular heat shock proteins are involved in cell-cell communication as well as immune and inflammatory processes.Hsp90 promotes cell survival, migration, inflammation and angiogenesis, and is therefore considered a promising target for cancer therapy.This led to the development of specific HSP90 inhibitors.More recently, these inhibitors have also been tested in diabetic animals.The use of the HSP90 inhibitor 17-DMAG significantly reduced atherosclerotic lesions and induced a more stable plaque phenotype in a mouse model with hyperglycemia and hyperlipidemia.Hsp90 is upregulated in human carotid atherosclerotic plaques (especially in unstable areas of plaques) and in patients' serums, triggering autoimmune antibodies against Hsp90 in patients.Is HSP90 also present in serum of patients with diabetic peripheral arterial disease?Is there a relationship between secretory heat shock protein 90 and arterial disease?The study that HSP90 may be involved in the molecular mechanism of vascular endothelial barrier function impairment in diabetes will provide a new target for the early serological diagnosis and treatment of diabetic vascular disease.The aim of this study was to investigate the relationship between the degree of vascular disease and serum heat shock protein 90 in patients with type 2 diabetes.The study was divided into three groups: diabetic without PAD group, diabetic with PAD group and diabetic foot group.According to the degree of peripheral artery disease, the patients were divided into three groups, and the content of heat shock protein 90 in serum of the patients was detected.To analyze the correlation between the degree of peripheral arterial disease and the content of heat shock protein 90 in serum.

DETAILED DESCRIPTION:
Diabetic foot disease with a global incidence of about 6% is one of the most serious complications of diabetes, which brings great pain and economic burden to patients.In China, the incidence rate is 8.1%, and the amputation rate is 7.3%. Every year, more than 1 million diabetic patients have amputations, ranking first among non-traumatic amputations.According to the American Diabetes Association (ADA), the incidence of Peripheral Arterial Disease (PAD) in diabetic patients is twice that of non-diabetic patients, and the resulting lower limb ischemia is the main cause of the high mortality and disability rate of diabetic foot.According to the International Working Group on Diabetic Foot (IWGDF), about 50% patients with diabetic foot disease are complicated with PAD, and the degree of vascular stenosis is closely related to the prognosis.Severe limb ischemia is a higher cause of diabetic foot ulcer in China than in western countries.Atherosclerosis is the main pathological change of diabetic peripheral artery disease, and endothelial injury is the initial link of atherosclerosis.Heat shock protein 90 (HSP90) is a kind of important heat stress protein, which accounts for about 2-3% of the total protein in cells.It is involved in the correct folding and activation of intracellular proteins.Although Hsp90 is primarily involved in intracellular protective mechanisms, they can also be exposed to the plasma membrane and released in the extracellular space, resulting in detectable levels of Hsp90 in the blood.Extracellular heat shock proteins are involved in cell-cell communication as well as immune and inflammatory processes.Hsp90 promotes cell survival, migration, inflammation and angiogenesis, and is therefore considered a promising target for cancer therapy.This led to the development of specific HSP90 inhibitors.More recently, these inhibitors have also been tested in diabetic animals.The use of the HSP90 inhibitor 17-DMAG significantly reduced atherosclerotic lesions and induced a more stable plaque phenotype in a mouse model with hyperglycemia and hyperlipidemia.Hsp90 is upregulated in human carotid atherosclerotic plaques (especially in unstable areas of plaques) and in patients' serums, triggering autoimmune antibodies against Hsp90 in patients.Is HSP90 also present in serum of patients with diabetic peripheral arterial disease?Is there a relationship between secretory heat shock protein 90 and arterial disease?The study that HSP90 may be involved in the molecular mechanism of vascular endothelial barrier function impairment in diabetes will provide a new target for the early serological diagnosis and treatment of diabetic vascular disease.The aim of this study was to investigate the relationship between the degree of vascular disease and serum heat shock protein 90 in patients with type 2 diabetes.The study was divided into three groups: diabetic without PAD group, diabetic with PAD group and diabetic foot group.According to the degree of peripheral artery disease, the patients were divided into three groups, and the content of heat shock protein 90 in serum of the patients was detected.To analyze the correlation between the degree of peripheral arterial disease and the content of heat shock protein 90 in serum.

1. Serum collection: the nurses collected the patients' fasting blood at 6:00 am in accordance with the routine blood collection procedures: 1 tube of procoagulant blood and 1 tube of anticoagulant blood were collected, each tube was no less than 3ml of blood;Store in a 4-degree refrigerator for disposal.
2. Collection of serum and plasma: the blood samples collected by the nurse were placed in a centrifuge, centrifuged at 3000 RPM for 15 minutes, and then the supernatant was collected.
3. Laboratory test: the collected serum or plasma were quantitatively tested by HSP90 ELISA, and the results were analyzed.The remaining serum or plasma was stored in a negative 80 refrigerator.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for diabetes: using WHO1999 diabetes diagnostic criteria, that is, (1) having diabetes symptoms (polyuria, polydipsia, and unexplained weight loss), and random (any time after meal) plasma glucose ≥11.1mmol/L(200mg/ dL);(2), or fasting (fasting for at least 8 hours) plasma glucose ≥7.0mmol/L(126mg/ dL);(3), or OGTT 2 hours plasma glucose ≥11.1mmol/L(200mg/ dL)
2. Inclusion criteria of the diabetes PAD group: patients diagnosed as T2DM according to the above-mentioned diagnostic criteria for diabetes, and with (1) symptoms and signs of atherosclerotic occlusion (intermittent claudication, resting pain, reduced or absent pulsation of dorsal foot artery, etc.);(2) Ankle-brachial arterial pressure index (ABI) ≤0.9;Toe brachial artery pressure index (TBI) ≤0.70;There was no three-phase pulse pattern of foot artery.Transcutaneous partial oxygen pressure (TcPO2) <30mmHg;(3) Evidence of atherosclerosis, atherosclerotic plaques, arterial stenosis or obstruction in carotid and/or lower extremity major arteries found by vascular color Doppler ultrasound.
3. Inclusion criteria for the diabetic foot group caused by PAD: the presence of infection, ulcer and/or deep tissue destruction of the foot was confirmed according to the above diagnostic criteria of diabetic PAD.
4. Agree to participate in the study and data collection, and sign the informed consent.

Exclusion Criteria:

-

1. Diabetic ketoacidosis or hyperosmolar state occurs within 30 days; Diabetic coma in 2 or 3 months, or severe hypoglycemia in nearly 1 month; 3. Diseases of tumor, immune system and hematopoietic system; 4. Other types of diabetes 5. Less than 40 years old

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 cases, 50 cases in each group.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Heat shock protein 90 | In December 2020
  The serum heat shock protein 90 was detected

CONTACTS AND LOCATIONS:
Overall Officials: Mengchen Zou, Principal Investigator — labor relations
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding X, Meng C, Dong H, Zhang S, Zhou H, Tan W, Huang L, He A, Li J, Huang J, Li W, Zou F, Zou M. Extracellular Hsp90alpha, which participates in vascular inflammation, is a novel serum predictor of atherosclerosis in type 2 diabetes. BMJ Open Diabetes Res Care. 2022 Jan;10(1):e002579. doi: 10.1136/bmjdrc-2021-002579. PMID 35091448

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT04787770/Prot_ICF_000.pdf